CLINICAL TRIAL: NCT00587145
Title: Phase II Study of Perioperative S-1 Plus Docetaxel in Patients With Localized Advanced Gastric Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Sook Ryun Park, M.D., National Cancer Center, Korea
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCCTS-06-190; 82-31-920-1609
Record Dates: First submitted 2007-12-21; First posted 2008-01-07 (Estimated); Last update posted 2008-01-07 (Estimated); Status verified 2007-12

CONDITIONS: Stomach Neoplasms
Keywords: Stomach Neoplasms; Secondary; Combination chemotherapy; S-1; Docetaxel; oxaliplatin
MeSH Terms: conditions — Stomach Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: S-1,Docetaxel — * S-1 80 mg/m2/day every 12-h p.o. on days 1(evening)-15 (morning)
  * Docetaxel 35 mg/m2 mixed in d5w 250 ml iv over 60-min on days 1 and 8

SUMMARY:
This study is an open-label, single center, and a single arm phase II study to evaluate the clinical response and safety of perioperative S-1 plus docetaxel. Perioperative chemotherapy is composed of 3 cycles of preoperative S-1/docetaxel and 3 cycles of postoperative S-1/docetaxel.Chemotherapy regimen:

* S-1 80 mg/m2/day every 12-h p.o. on days 1(evening)-15 (morning)
* Docetaxel 35 mg/m2 mixed in d5w 250 ml iv over 60-min on days 1 and 8

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed localized gastric adenocarcinoma as defined by CT stage III and IV (M0) (but not N3, which is metastatic node in WHO TNM classification), according to Japanese TNM classification system
2. No distant metastatic disease in laparoscopy
3. Age: 18-70 years
4. Eastern Cooperative Oncology Group (ECOG) performance status 0-1
5. Disease status must be that of measurable disease as defined by RECIST: Measurable lesions: lesions that can be accurately measured in at least one dimension by abdominal CT, if the longest diameter to be recorded is at least 10 mm with spiral CT
6. Adequate major organ function including the following: Hematopoietic function: WBC ³ 4,000/mm3, ANC ³ 1,500/mm3, Platelet ³ 100,000/mm3Hepatic function: serum bilirubin £ 1.5 mg/dl, AST/ALT levels £ 2.5 x UNLRenal function: serum creatinine £ 1.5 mg/dl
7. Patients should sign a written informed consent before study entry

Exclusion Criteria:

1. CT Stage I, II, M1 or N3, which is metastatic node in WHO TNM classification, according to Japanese TNM classification system
2. Prior chemotherapy or radiotherapy
3. Inadequate cardiovascular function:New York Heart Association class III or IV heart diseaseUnstable angina or myocardial infarction within the past 6 monthsHistory of significant ventricular arrhythmia requiring medication with antiarrhythmics or significant conduction system abnormality
4. Serious concurrent infection or nonmalignant illness that is uncontrolled or whose control may be jeopardized by complications of study therapy
5. Other malignancy within the past 3 years except non-melanomatous skin cancer or carcinoma in situ of the cervix
6. Psychiatric disorder that would preclude compliance
7. Pregnant, nursing women or patients with reproductive potential without contraception
8. Patients receiving a concomitant treatment with drugs interacting with S-1 such as flucytosine, phenytoin, or warfarin et al.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2006-05; Primary Completion 2009-03 (Estimated); Study Completion 2009-05 (Estimated)

PRIMARY OUTCOMES:
To evaluate the clinical responses to preoperative S-1 plus docetaxel | During chemotherapy

SECONDARY OUTCOMES:
the clinical downstaging,the pathologic responses, toxicity profile,the disease-free survival,overall survival,the effect of CYP2A6 genetic polymorphisms on the pharmacokinetics and the difference in pharmacokinetics between before and after gastrectomy | During study period

CONTACTS AND LOCATIONS:
Overall Officials: Sook Ryun Park, M.D, Principal Investigator — National Cancer Center, Korea
Locations (1):
- National Cancer Center Korea, Goyang-si, Gyeonggi-do, South Korea